CLINICAL TRIAL: NCT06229665
Title: An Open-Label, Prospective, Multi-Center Extension Study to Assess the Long-Term Safety and Efficacy of Photobiomodulation (PBM) in Subjects With Dry Age-Related Macular Degeneration (AMD) (LIGHTSITE IIIB)
Brief Title: Study of Photobiomodulation to Treat Dry Age-Related Macular Degeneration (LIGHTSITEIIIB)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: LumiThera, Inc. (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP010
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-04

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: dry age-related macular degeneration; photobiomodulation

STUDY DESIGN:
Intervention Model Description: Valeda Light Delivery System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Photobiomodulation (PBM) (Experimental): The Valeda Light Delivery System will deliver two alternating and sequential treatments of 590 nm and 850 nm for 35 seconds, or a total of 70 seconds; and 660 nm for 90 seconds, or a total of 180 seconds.
  Interventions: Device: Valeda Light Delivery System

INTERVENTIONS:
Device: Valeda Light Delivery System — The Valeda Light Delivery System will deliver two alternating and sequential treatments of 590 nm and 850 nm for 35 seconds, or a total of 70 seconds; and 660 nm for 90 seconds, or a total of 180 seconds.

SUMMARY:
This study is an open-label, prospective, multi-center extension study on the continued use of photobiomodulation (PBM) in subjects with dry age-related macular degeneration (AMD) that participated in the CSP005 LIGHTSITE III study.

DETAILED DESCRIPTION:
This study is an open-label, prospective, multi-center study on the use of PBM as a treatment for visual impairment in subjects with dry AMD. Subjects diagnosed with dry AMD who meet all inclusion criteria and have none of the exclusion criteria will be eligible to participate in this clinical study. All subjects will be treated with the Valeda Light Delivery System and will receive PBM treatment for a total of 9 treatments over a three to five-week period (3 times per week for 3 weeks is preferable). There will be a re-treatment period starting at the 4-month time point to include 9 additional treatment visits, to be repeated again at 8 months and 12 months. LumiThera will use settings for the 3 wavelengths that were used in the CSP005 study. The subject population for this study will consist of all subjects that completed the CSP005 study, meet the inclusion/exclusion criteria for the CSP010 study, are interested in study participation and have signed the Informed Consent Form.

ELIGIBILITY:
Entry Criteria: Inclusion Criteria (each eye qualifies for the study independently):

1. Participation in and completion of LIGHTSITE III study.
2. Eye was randomized in LIGTHTSITE III study or diagnosis of dry AMD as defined by the presence of the following: Drusen that are intermediate in size or larger (63 μm or larger in diameter) with at least a few (3) being regular drusen and not pseudodrusen and/or geographic atrophy (GA) visible on two of the following: color fundus images, OCT and/or FAF. The reading center will confirm criteria for NEW EYES only (i.e., those not randomized in LIGHTSITE III) with one of the following: 1) LIGHTSITE IIIB Screening Visit images (Screening visit only performed if there are >90 days between LIGHTSITE III Mo 24 visit and the start of the LIGHTSITE IIIB study) or 2) LIGHTSITE III Mo 24 images (if <90 days passes between LIGHTSITE III Mo 24 and the start of the LIGHTSITE IIIB study).
3. Able to communicate well with the Investigator and able to understand and comply with the requirements of the study
4. Informed of the nature of this study and has provided written, informed consent in accordance with institutional, local and national regulatory guidelines

Exclusion Criteria (each eye qualifies for the study independently):

1. Current or history of neovascular maculopathy that includes any of the following (to be confirmed by the reading center):

   1. Choroidal neovascularization (CNV) defined as pathologic angiogenesis originating from the choroidal vasculature that extends through a defect in Bruch's membrane
   2. Serous and/or hemorrhagic detachment of the neurosensory retina or retinal pigment epithelial (RPE)
   3. Retinal hard exudates (a secondary phenomenon resulting from chronic intravascular leakage)
   4. Subretinal and sub-RPE fibrovascular proliferation
   5. Disciform scar (subretinal fibrosis)
2. Media opacities, including cataracts, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require cataract surgery in the study eye in the next 12 months.
3. Posterior capsule opacification, which might interfere with visual acuity or imaging in the study eye(s). Subjects should not be entered if there is likelihood that they will require surgery in the study eye in the next 12 months.
4. Invasive eye surgery (e.g. cataract, capsulotomy) on a qualifying eye within three months prior to Baseline
5. Ocular disorder or disease that partially or completely obstructs the pupil (e.g. posterior synechia in uveitis)
6. Visually significant disease in any ocular structure apart from dry AMD (e.g. diabetic macular edema, glaucoma (using >2 eye drop medications, uncontrolled IOP and/or central/paracentral visual field loss), glaucoma surgery, active uveitis, active vitreous disease, intraocular tumor, retinal vascular diseases)
7. Ocular disorder or disease other than dry AMD that could cause drusen (glomerulonephritis Type 2, Autosomal dominant drusen), GA (North Carolina dystrophy) or mitochondrial diseases (parafoveal petaloid GA, Stargardt disease)
8. Presence or history of disease or condition affecting functional vision without obvious structural abnormalities (e.g. amblyopia, stroke, nystagmus)
9. Serious medical illness that will prevent the subject from performing study activities (including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease) or, in the judgement of the Investigator, is likely to require surgical intervention or hospitalization at any point during the study
10. Presence of or history of malignancy within the past 3 years other than non-melanoma skin or squamous cell cancer or cervical carcinoma in-situ
11. Is non-ambulatory
12. Presence or history of known light sensitivity to yellow light, red light, or near infrared radiation (NIR), or if they have a history of light activated CNS disorders (e.g. epilepsy, migraine)
13. Use of any photosensitizing agent (e.g. topicals, injectables, oral) activated by the Valeda Light Delivery System wavelengths within 30 days of treatment without consulting subject's physician
14. History of drug, alcohol or substance abuse within 3 months prior to Baseline
15. Participation in any other clinical study at time of Baseline, or has received an investigational drug or treatment with an investigational device within 3 months prior to Baseline
16. If on any anti-oxidant or vitamin Age-Related Eye Disease Study (AREDS) supplement for dry AMD, has not been stabilized for a minimum of 1 month prior to Baseline. Subjects are considered to be stable if they are taking the AREDS supplements consistently as prescribed by their treating doctor.
17. Has received Low Vision Rehab/Therapy within 30 days prior to Baseline or intends to receive during the study
18. Has an open sore(s) that may come in contact with the Valeda System, has periorbital skin erythema or is prone to such conditions with exposure to light.
19. In the opinion of the Investigator, is unlikely to comply with the study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Early Treatment Diabetic Retinopathy Study (ETDRS) Best-Corrected Visual Acuity (BCVA) | 12 months
  Mean change from baseline in BCVA.

SECONDARY OUTCOMES:
Low Luminance BCVA | 12 months
  Mean change from baseline in the LLBVCA.
Contrast Seensitivity | 12 months
  Mean change from baseline (pre-treatment) in contrast sensitivity at 80 cm and 120 cm.
Geographic Atrophy (GA) | 12 months
  Number of new onset GA

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Stanford University, Palo Alto, California
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - New York Ear and Eye Infirmary, New York, New York
  - Gulf Coast Eye Institute, McAllen, Texas
  - Retina Center Northwest, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No